CLINICAL TRIAL: NCT06439836
Title: Phase 1 Trial of CA-4948 in Combination With Pembrolizumab to Overcome Resistance to PD-1/PD-L1 Blockade in Metastatic Urothelial Cancer
Brief Title: Pembrolizumab Plus CA-4948 for the Treatment of Patients With Progressive Metastatic Urothelial Cancer Despite Prior Immunotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-04436; NCI-2024-04436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10636 (Other: NY021 Mount Sinai Hospital); 10636 (Other: CTEP)
Record Dates: First submitted 2024-05-31; First posted 2024-06-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Urothelial Carcinoma; Unresectable Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Biopsy; Specimen Handling; CA-4948; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CA-4948, pembrolizumab) (Experimental): Patients receive CA-4948 orally PO BID on days 1-21 and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, CT, MRI, or PET throughout the study. Additionally, patients may undergo a tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Emavusertib; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Emavusertib — Given PO
  Other Names: AU 4948; AU-4948; CA 4948; CA-4948; CA4948; Interleukin-1 Receptor-associated Kinase 4 Inhibitor CA-4948; IRAK4 Inhibitor CA-4948
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase I trial tests the safety, side effects, best dose, and effectiveness of emavusertib (CA-4948) in combination with pembrolizumab in treating patients with urothelial cancer that has spread from where it first started to other places in the body (metastatic) and that has a resistance to PD-1/PD-L1 immune checkpoint inhibitors. CA-4948, a kinase inhibitor, may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving CA-4948 in combination with pembrolizumab may be safe, tolerable and/or effective in treating patients with metastatic urothelial cancer that is resistant to PD-1/PD-L1 immune checkpoint inhibitors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose of the combination of CA-4948 plus pembrolizumab in patients with immune checkpoint blockade (ICB)-resistant metastatic urothelial cancer (Dose Escalation Cohort).

II. To determine the safety of the combination of CA-4948 plus pembrolizumab in patients with ICB-resistant metastatic urothelial cancer (Dose Escalation Cohort and Dose Expansion Cohort).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To measure the objective response (complete response [CR] or partial response [PR]) as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at 9 weeks and the best overall response (CR or PR) as defined by RECIST 1.1 at any time while on study.

III. To determine progression-free survival, overall survival, and duration of response.

IV. To assess whether CA-4948 plus pembrolizumab leads to on-treatment increases in 2IR scores (as defined by ribonucleic acid [RNA] sequencing) in paired tumor biopsies.

EXPLORATORY OBJECTIVES:

I. To assess the clinical benefit rate with pembrolizumab plus CA-4948 therapy. II. To assess the "C-reactive protein (CRP) response rate" as defined by the proportion of patients achieving a ≥ 1.5 fold reduction in CRP at 9 weeks.

III. To explore the association between the 2IR score as defined by bulk-ribonucleic acid (RNA) sequencing of pre-treatment tumor tissue and objective response rate, clinical benefit rate, progression-free survival, and/or overall survival.

IV. To explore whether CA-4948 plus pembrolizumab leads to on-treatment changes in the cellular and/or molecular composition of the tumor microenvironment (TME).

V. To explore the association between the quantity and spatial localization of SPP1+ monocytes-macrophages (MoMacs) defined by multiplex immunohistochemistry on pre-treatment tumor tissue and objective response rate, clinical benefit rate, progression-free survival, and/or overall survival.

VI. To explore the association between the cellular and molecular composition of the TME defined by spatial RNA sequencing on pre-treatment tumor tissue and objective response rate, clinical benefit rate, progression-free survival, and/or overall survival.

VII. To explore on-treatment changes in high-sensitivity (hs) CRP and cytokines and chemokines in peripheral blood and their association with objective response rate, clinical benefit rate, progression-free survival, and/or overall survival.

VIII. To explore the association between PD-L1 expression on pre-treatment tumor tissue and objective response rate, clinical benefit rate, progression-free survival, and/or overall survival.

IX. To explore the association between the CXCL9:SPP1 ratio as defined by bulk-RNA sequencing of pre-treatment tumor tissue and objective response rate, clinical benefit rate, progression-free survival, and/or overall survival.

X. To assess whether CA-4948 plus pembrolizumab leads to on-treatment increases in the CXCL9:SPP1 ratio (as defined by RNA sequencing) in paired tumor biopsies.

OUTLINE: This is a dose-escalation study of CA-4948 in combination with pembrolizumab followed by a dose-expansion study.

Patients receive CA-4948 orally (PO) twice daily (BID) on days 1-21 and pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection, computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) throughout the study. Additionally, patients may undergo a tumor biopsy on study.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed urothelial cancer that is metastatic or unresectable and must have had the prior treatments outlined
* Age ≥ 18 years

  * Because no dosing or adverse event data are currently available on the use of CA-4948 in combination with pembrolizumab in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%) within 28 days prior to registration
* Leukocytes ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L

  * Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin (≥ approximately 3 months)
* Creatine phosphokinase (CPK) < grade (Gr) 2 ( </= 2.5 upper limit of normal [ULN])
* Creatinine < 1.5 × institutional ULN or creatinine clearance of ≥ 30 mL/min for patient with creatine levels ≥ 1.5 x institutional ULN

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 3 x ULN
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x ULN
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Ability to provide at least 20 unstained slides or formalin-fixed paraffin-embedded (FFPE) block plus 1 hematoxylin and eosin (H&E) slide from prior archival invasive urothelial cancer specimen (and/or ability to undergo baseline tumor biopsy in patients in the expansion cohort)
* Measurable metastatic or unresectable disease
* Must have received prior treatment with a PD-1 or PD-L1 inhibitor
* Must have received at least one of the following (may have been administered concurrently or sequentially with PD-1/PD-L1 inhibitor):

  * Platinum-based chemotherapy
  * Enfortumab vedotin
* Primary resistance to PD-1/PD-L1 blockade as defined by Society for Immunotherapy of Cancer (SITC) consensus definitions:

  * For patients who received single-agent PD-1/PD-L1 blockade in the adjuvant setting:

    * Must have received ≥ 6 weeks of treatment with PD-1/PD-L1 blockade
    * Recurrence while on treatment or within ≤ 3 months after completion of therapy
  * For patients who received single-agent PD-1/PD-L1 blockade in the metastatic setting:

    * Must have received ≥ 6 weeks of treatment with PD-1/PD-L1 blockade
    * Progression within ≤ 6 months of initiating treatment with single-agent PD-1/PD-L1 blockade with best response of stable disease
  * For patients who received single-agent PD-1/PD-L1 blockade in the switch-maintenance setting:

    * Must have received ≥ 6 weeks of treatment with PD-1/PD-L1 blockade
    * Progression within ≤ 6 months of initiating treatment with single-agent PD-1/PD-L1 blockade
  * For patients who received an antibody-drug conjugate or cytotoxic chemotherapy plus PD-1/PD-L1 blockade combination

    * Must have received ≥ 6 weeks of treatment with PD-1/PD-L1 blockade
    * Progression within ≤ 12 months of initiating treatment
  * An eligibility form will be developed to include documentation of the dates of prior PD-1/PD-L1 blockade and a redacted radiology report confirming best response of stable disease for < 6 months or progressive disease)
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Female patients of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Patients who have received messenger ribonucleic acid (mRNA) coronavirus disease 2019 (COVID-19) and influenza vaccines will be allowed
* Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either magnetic resonance imaging [MRI] or computed tomography [CT] scan, for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patients should be willing and able to swallow pills
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) Note: Patients with grade ≤ 2 neuropathy or grade ≤ 2 alopecia are an exception to this criterion and may qualify for the study. Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Grade ≥ 3 immune related adverse event with prior PD-1/PD-L1 blockade
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CA-4948 and/or pembrolizumab
* Patients with uncontrolled intercurrent illness, including but not limited to interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia that would limit compliance with study requirements
* Patients who are receiving any other investigational agents
* Patients with carcinomatous meningitis
* Patients with malabsorption syndrome or other conditions that would interfere with intestinal absorption
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has received a live vaccine within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted
* Pregnant women are excluded from this study because pembrolizumab is a monoclonal antibody with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab, breastfeeding should be discontinued if the mother is treated with pembrolizumab. These potential risks may also apply to other agents used in this study
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] RNA [qualitative] is detected)
* Has a known history of active tuberculosis (TB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) | Up to completion of cycle 1
  Adverse events (AEs) will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Occurrence of DLTs along with count and percentage of subjects experiencing DLTs will be summarized. Safety of the combination regimen will be summarized by the number of adverse events as well as by the number and percentage of subjects experiencing the adverse events in both dose escalation and expansion cohorts. The safety summary will include count and percentage for overall and by AE type, seriousness, severity, attribution, anticipated or not. Furthermore, toxicity index will be calculated as a summary index for each patient to summarize multiple AEs.
Recommended phase 2 dose (RP2D) | Up to completion of cycle 1
  The RP2D may be determined to be the highest dose level, the maximum tolerated dose, or it may be a lower dose based on the consensus of the investigators, Cancer Therapy Evaluation Program and pharmaceutical company collaborators.
Incidence of AEs | Up to 30 days after last dose of study treatment
  AEs will be graded using NCI CTCAE v 5.0. Safety will be summarized by the number of AEs as well as by the number and percentage of subjects experiencing the AEs in both the dose escalation and dose expansion phases of the study. The safety summary will include count and percentage for overall and by AE type, seriousness, severity, attribution, anticipated or not. Toxicity will be calculated as a summary index for each patient to summarize multiple AEs.

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 9 weeks
  ORR will be defined as the proportion of patients achieving a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria at 9 weeks. The number of confirmed responses will be reported along with a corresponding two-sided 95% Wilson confidence interval (CI) and p-value will be reported from Binomial exact test.
Progression-free survival (PFS) | At initial treatment to progression or death up to 2 years after last dose of study treatment
  PFS will be defined as the time from initial treatment to any progression or death from any cause, whichever occurs first. Kaplan-Meier estimates of median PFS time will be presented together with two-sided 95% CIs calculated according to Brookmeyer and Crowley. The frequency (number and percentage) of participants with an event (progression or death) and censoring reasons will be presented (alive, withdrawal of consent, lost to follow-up).
Overall survival (OS) | At start of study treatment to death up to 2 years after last dose of study treatment
  OS will be defined as the duration from the first date of study treatment to the date of death. Kaplan-Meyer estimates of median OS will be presented together with two-sided 95% CIs calculated according to Brookmeyer and Crowley. the frequency of participants with an event and censoring reasons will be presented.
Duration of response (DOR) | At first response to progression or death up to 2 years after last dose of study treatment
  DOR will be defined as the time from date of the first documentation of response to the first documentation of progression of disease or death due to any cause in the absence of documented progression of disease. Kaplan-Meier estimates of median DOR time will be presented together with two-sided 95% CIs calculated according to Brookmeyer and Crowley. The frequency of participants with an event and censoring reasons will be presented.
2IR scores | At baseline and up to 2 years after last dose of study treatment
  The 2IR score will be calculated using the mean expression levels of the adaptive immune response and pro-tumorigenic inflammation gene signatures from the baseline and on-treatment transcriptome profile derived for each subject. A paired t-test will be used to test whether there is an increase in 2IR score from baseline to on-treatment time points. Univariable logistic regression models will be fitted for response variables with either 2IR score at baseline and change in 2IR score as continuous covariates. Proportional hazard (PH) Cox regression models for PFS and OS will also be fitted with 2IR score either at baseline or as time-dependent continuous covariates.

OTHER OUTCOMES:
Clinical benefit rate (CBR) | At 9 weeks
  CBR will be defined as the proportion of patients achieving a CR or PR per RECIST 1.1 criteria at 9 weeks or stable disease at 9 weeks accompanied by a 1.5 or greater reduction in hrCRP. CBR will be reported along with a corresponding two-sided 95% Wilson CI and p-value will be reported from Binomial exact test.
High-sensitivity C-reactive protein (hsCRP) | At 9 weeks
  CRP response rate will be defined as achieving a ≥ 1.5 fold reduction in CRP at 9 weeks. The CRP response rate will be reported along with a corresponding two-sided 95% Wilson CI and p-value will be reported from Binomial exact test. Linear mixed models will also be fitted for comparisons between patients achieving and not achieving an objective response and between patients achieving and not achieving clinical benefit. Random effects with autoregressive model of order 1 will be incorporated to describe the correlation of repeated measures. Univariable PH Cox regression models for PFS and OS will also be fitted with hsCRP levels either at baseline or as a time-dependent continuous covariate.
Cyotkines and chemokines | At baseline and up to 2 years after last dose of study treatment
  Linear mixed models will also be used for comparisons between patients achieving and not achieving an objective response and between patients achieving and not achieving clinical benefit. Random effects with autoregressive model of order 1 will be incorporated to describe the correlation of repeated measures. Residual plots will be used to check model assumptions. Univariable PH Cox regression models for PFS and OS will also be fitted with cytokine and chemokine levels either at baseline or as time-dependent continuous covariates. Schoenfeld residuals will be used to check PH assumption. P-values will be adjusted by false discovery rate of 5%.
Multiplex immunohistochemistry markers | At baseline and up to 2 years after last dose of study treatment
  A paired t-test will be used to test whether there are a reduction of SPP1+ MoMacs and an increase in intra-tumoral T cells from baseline to on-treatment time points. Univariable logistic regression models will be fitted for ORR and CBR as response variables with either marker levels at baseline or change in marker levels as continuous covariates. PH Cox regression models for PFS and OS will also be fitted with marker levels either at baseline or as time-dependent continuous covariates. Schoenfeld residuals will be used to check PH assumption. P-values will be adjusted by false discovery rate of 5%.
PD-L1 expression | Up to 2 years after last dose of study treatment
  Univariable logistic regression models will be fitted for ORR and CBR as response variables with PD-L1 expression as continuous covariate. Univariable PH Cox regression models for PFS and OS will be fitted with PD-L1 expression as continuous covariate. Schoenfeld residuals will be used to check PH assumption.
Tumor microenvironment (TME) markers | At baseline and up to 2 years after last dose of study treatment
  A paired t-test will be used to test whether there are a decrease in SPP1+ CD68+ cells and an increase in C1QC+ CD68+ cells from baseline to on-treatment time points. Univariable logistic regression models will be fitted for ORR and CBR as response variables with either TME markers at baseline or change in TME marker levels as continuous covariates. PH Cox regression models for PFS and OS will be fitted with TME markers either at baseline or as time-dependent continuous covariates. Schoenfeld residuals will be used to check PH assumption. P-values will be adjusted by false discovery rate of 5%.
Cytometry by time of flight | At week 1 of cycles 1-3
  Will be analyzed using state of the art techniques developed at National Institute of Health and Mount Sinai focused on modeling variance and cellular abundance of these cell populations. The hierarchical nature of the classification and identification of cell types will allow to characterize and identify what populations are affected by treatment and associated with response in the periphery, in contrast with the data obtained at the tumor site (locally), which is identified with spatial assays.
Extracellular vesicles and particles (EVPs) | At week 1 of cycles 1-3
  Will be analyzed using linear mixed models for longitudinal comparisons, univariable logistic regression for associations with ORR and CBR, and proportional hazards Cox models (including time-dependent covariates) for PFS and OS. Model assumptions will be evaluated using residual diagnostics, including Schoenfeld residuals for PH models. False discovery rate adjustment at 5% will be applied for multiple testing correction. EVP-derived molecular signatures (also known as the secretome) may provide complementary, non-redundant insights beyond those captured by Olink, immunohistochemistry, and spatial transcriptomics, and may identify circulating surrogates of treatment response or resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Galsky, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (11):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm